CLINICAL TRIAL: NCT00898391
Title: Analysis of Circulating MYCN DNA in Serum Samples Obtained From Patients With Neuroblastoma
Brief Title: Study of DNA in Blood Samples From Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL07B1; NCI-2009-00686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-NB2006-10 (Other: Children's Oncology Group); NB2006-10 (Other: Children's Oncology Group); ANBL07B1 (Other: CTEP)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Disseminated Neuroblastoma; Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Polymerase Chain Reaction; Electrophoresis, Polyacrylamide Gel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative: Circulating DNA is extracted from serum. PCR amplification of MYCN is performed and analyzed by agarose gel electrophoresis. Real-time quantitative PCR is also performed.
  Interventions: Other: laboratory biomarker analysis; Genetic: polymerase chain reaction; Genetic: polyacrylamide gel electrophoresis; Genetic: DNA analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: polyacrylamide gel electrophoresis — Correlative studies
  Other Names: electrophoresis, polyacrylamide gel
Genetic: DNA analysis — Correlative studies

SUMMARY:
This research trial studies is deoxyribonucleic acid (DNA) in blood samples from patients with neuroblastoma. Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Perform in a blind study a multicentric study by analyzing serum from patients at diagnosis (with a known tumor v-myc avian myelocytomatosis viral oncogene neuroblastoma derived homolog (MYCN) status determined in the Children's Oncology Group [COG] reference lab), in order to confirm our previous data and to define the most appropriate MYCN/control ratio cutoff capable of determining positive and negative cases.

II. Define the limits of the procedure in non-metastatic patients and in those with reduced tumor burden (International Neuroblastoma Staging System [INSS] stage 1 and 2).

OUTLINE:

Circulating DNA is extracted from serum. Polymerase chain reaction (PCR) amplification of MYCN is performed and analyzed by agarose gel electrophoresis. Real-time quantitative PCR is also performed.

ELIGIBILITY:
Inclusion Criteria:

* Serum samples from neuroblastoma (NB) patients obtained through the COG (and legacy Children's Cancer Group [CCG]/Pediatric Oncology Group [POG] Biology Studies)

  * The MYCN status on corresponding tumors have been determined using standard techniques; the panel of samples must be obtained from NB patients with and without MYCN amplification tumors
* Cases will be drawn from clinical subsets at greatest likelihood to benefit from this testing ability, stage 1 and 2 NBs (both infants and toddlers), stage 4 patients under 18 months of age, and 4S patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neuroblastoma treated at a COG participating site.
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2007-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Most appropriate MYCN/control ratio cutoff capable of determining positive and negative cases of neuroblastoma assessed by PCR | Up to 6 months
Limits of the procedure in non-metastatic patients and in those with reduced tumor burden | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hogarty, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States